CLINICAL TRIAL: NCT05536193
Title: Efficacy and Safety of Topical Metformin Emulgel Versus Salicylic Acid Peeling in Treatment of Acne Vulgaris: A Split Face Study
Brief Title: Topical Metformin Emulgel VS Salicylic Acid Peeling in Treatment of Acne Vulgaris
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ola Ahmed Elminshawy, Principal Investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMEVSSA
Record Dates: First submitted 2022-09-07; First posted 2022-09-10 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Salicylic Acid

STUDY DESIGN:
Intervention Model Description: Patients will use salicylic acid 30% peeling on the right side of the face and topical metformin emulgel on the left side
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Topical Metformin Emulgel and salicylic acid (Experimental)
  Interventions: Drug: Topical Metformin Emulgel and salicylic acid; Diagnostic Test: Insulin- Like growth factor (ILGF-1)

INTERVENTIONS:
Drug: Topical Metformin Emulgel and salicylic acid — Combination Product: Topical metformin emulgel topical metformin emulgel will be used on the left side of the face twice daily (home use).
  Procedure/Surgery: Salicylic acid Patients will have salicylic acid 30% peeling on the right side of the face as a peeling session every two weeks. Sessions will be done by well trained physician.
  Other Names:
  • 2-hydroxybenzoic acid
Diagnostic Test: Insulin- Like growth factor (ILGF-1) — 3 ml blood for serum sample for estimation of Insulin- Like growth factor (ILGF-1) by ELISA kit will be taken from every patient before and after use of topical metformin.

SUMMARY:
Acne Vulgaris (AV ) is a common skin disorder worldwide, affecting all ages and races, considered as a long term chronic inflammatory disease of the skin.It affects nearly 85% of adolescents and about 30% of adults which is known as post- adolescent acne that often occurs in individuals aged 25 years or older particularly women.

Acne lesions, which may be papules, pustules, or nodules commonly affecting face, chest and back therefore acne patients may suffer from emotional distress due to its chronicity and potential outcomes which include physical scars and persistent hyperpigmentation.

The pathophysiology of AV involves four factors: abnormal follicular keratinization, hyperseborrhea, Cutibacterium acnes proliferation in the pilosebaceous unit and inflammatory mediators released into the skin.

Diet is considered to be one of the main factors influencing the induction and aggravation of acne, though this is still debatable. Previous researches have focused on glycemic load, and hyperinsulinemia which lead to an increase in the concentration of insulin-like growth factor (IGF-1), which has been reported to affect androgen metabolism and lipogenesis Additionally, IGF-1 has been shown to upregulate inflammatory cytokines. A correlation between the severity of acne and the level of serum IGF-1 has also been reported. Previous clinical studies showed that a low glycemic diet can decrease both the size of the sebaceous gland and the number of inflammatory lesions

DETAILED DESCRIPTION:
Several treatment modalities have been used to treat AV. Topical therapies include antibiotics, azelaic acid, benzoyl peroxide, and retinoids. Systemic treatments include antibiotics, hormonal therapy, and isotretinoin in addition to physical modalities as chemical peeling .

Chemical peeling is a safe, efficacious, and cost-effective procedure for treating various skin disorders and for enhancing cosmetic appearance. The principle of peeling involves controlled chemical injury to the skin in order to promote it to rejuvenate, leading to smoothening of the skin and improvement of its surface texture .

As patients become more concerned about the risks and side-effects of acne medications such as antibiotics and isotretinoin, other options are needed .

Metformin is an oral antihyperglycemic agent often used to treat overweight type 2 diabetic patients. It decreases hepatic glucose output and increases glucose utilization by muscles and adipocytes by increasing insulin sensitivity .

Notably, metformin has been shown to suppress the mammalian target of rapamycin complex (mTORC1) activity . mTORC, also known as the mechanistic target of rapamycin, is a central cell growth regulating kinase that forms large molecular complexes in all eukaryotic cells. Rapamycin is an mTORC1-specific inhibitor, which complexes with the FK506-binding 12 kDa protein (FKBP12). Rapamycin analogs have been used clinically to treat a number of human diseases, including cancer. A wide range of both extra- and intracellular signals, including growth factors, nutrient status and stress conditions, have been shown to regulate mTORC1 to control cell growth .

Hence, it is plausible that metformin through inhibition of mTORC1 improves acne as AV is one of the mechanistic target of rapamycin complex 1 (mTORC1)-driven diseases. Moreover, metformin has been suggested for the treatment of other insulin resistant-related skin disorders such as hirsutism, hidradenitis suppurativa, and acanthosis nigricans .

In order to get a benefit from the anti-inflammatory effect of metformin on the skin, the best option is to enhance its dermal effects, therefore, its side effects will be less through the topical administration route .

Actually, by applying a topical form of this drug on acne spots, mTORC1 over activation in skin cells can be inhibited which leads to disappearance of acne spots .

Salicylic acid (SA) is a safe and efficacious peeling agent for a number of dermatological and cosmetic problems, including acne vulgaris .

SA peels soften the stratum corneum and cause skin shedding by loosening the intracellular matrix and corneocyte connections which can lead to an improvement in non-inflammatory comedones . Also, SA inhibits the arachidonic acid cascade leading to a decrease in inflammatory lesions .

In our study, we chose the emulgel formulation as a topical metformin form to increase the efficacy and absorption in treatment of AV. Emulgel used will be optimized for biocompatibility, consistency and chemical compatibility with metformin.

ELIGIBILITY:
Inclusion Criteria:

* Both males and females will be included.
* Patients older than 18 years of age.
* Patients with mild and moderate AV.
* Patients with Fitzpatrick skin type III, IV and V.

Exclusion Criteria:

* Severe acne.

  * Patients under treatment with contraceptive pills or received any kinds of systemic or topical acne medication in the last 2 months (isotretinoin, antibiotics, topical products) or corticosteroid, lithium, growth hormone, systemic metformin, vitamin B12, whey proteins, and estrogenic-progestogens.
  * History of hypertrophic/keloid scar formation.
  * Pregnancy and lactation.
  * Recurrent herpes infection.
  * Subjects with diseases that affect IGF-1 levels such as diabetes, metabolic syndrome, and acromegaly.
  * Conditions that affect liver or thyroid function, celiac disease and inflammatory bowel diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2022-09-10 (Estimated); Primary Completion 2023-09-10 (Estimated); Study Completion 2023-09-10 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the medications | 12 weeks
  by counting the number of inflammatory, non-inflammatory and total lesions at baseline and every 4 weeks during the treatment.
Evaluate effect of topical metformin on decreasing serum concentration of insulin-like growth factor 1 (IGF-1) | 12 weeks
  Evaluate effect of topical metformin on decreasing serum concentration of insulin-like growth factor 1 (IGF-1) by serum sample that will be taken from every patient before and after use of topical metformin.

SECONDARY OUTCOMES:
Assessment of tolerability | 12 weeks
  by interviewing the patients about any sign/symptom of adverse reactions (erythema, peeling, burning sensation, dryness and pruritus).
Assessment of patient satisfaction | 12 weeks
  by quartile grading system

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Titus S, Hodge J. Diagnosis and treatment of acne. Am Fam Physician. 2012 Oct 15;86(8):734-40. PMID 23062156
- [Background] Han XD, Oon HH, Goh CL. Epidemiology of post-adolescence acne and adolescence acne in Singapore: a 10-year retrospective and comparative study. J Eur Acad Dermatol Venereol. 2016 Oct;30(10):1790-1793. doi: 10.1111/jdv.13743. Epub 2016 Jul 12. PMID 27400809
- [Background] Hazarika N, Archana M. The Psychosocial Impact of Acne Vulgaris. Indian J Dermatol. 2016 Sep-Oct;61(5):515-20. doi: 10.4103/0019-5154.190102. PMID 27688440
- [Background] Williams HC, Dellavalle RP, Garner S. Acne vulgaris. Lancet. 2012 Jan 28;379(9813):361-72. doi: 10.1016/S0140-6736(11)60321-8. Epub 2011 Aug 29. PMID 21880356
- [Background] Kim H, Moon SY, Sohn MY, Lee WJ. Insulin-Like Growth Factor-1 Increases the Expression of Inflammatory Biomarkers and Sebum Production in Cultured Sebocytes. Ann Dermatol. 2017 Feb;29(1):20-25. doi: 10.5021/ad.2017.29.1.20. Epub 2017 Feb 3. PMID 28223742
- [Background] Kwon HH, Yoon JY, Hong JS, Jung JY, Park MS, Suh DH. Clinical and histological effect of a low glycaemic load diet in treatment of acne vulgaris in Korean patients: a randomized, controlled trial. Acta Derm Venereol. 2012 May;92(3):241-6. doi: 10.2340/00015555-1346. PMID 22678562
- [Background] Fox L, Csongradi C, Aucamp M, du Plessis J, Gerber M. Treatment Modalities for Acne. Molecules. 2016 Aug 13;21(8):1063. doi: 10.3390/molecules21081063. PMID 27529209
- [Background] Rendon MI, Berson DS, Cohen JL, Roberts WE, Starker I, Wang B. Evidence and considerations in the application of chemical peels in skin disorders and aesthetic resurfacing. J Clin Aesthet Dermatol. 2010 Jul;3(7):32-43. PMID 20725555
- [Background] Badr D, Kurban M, Abbas O. Metformin in dermatology: an overview. J Eur Acad Dermatol Venereol. 2013 Nov;27(11):1329-35. doi: 10.1111/jdv.12116. Epub 2013 Feb 26. PMID 23437788
- [Background] Yuan HX, Guan KL. Structural insights of mTOR complex 1. Cell Res. 2016 Mar;26(3):267-8. doi: 10.1038/cr.2016.10. Epub 2016 Jan 22. PMID 26794870
- [Background] Arif T. Salicylic acid as a peeling agent: a comprehensive review. Clin Cosmet Investig Dermatol. 2015 Aug 26;8:455-61. doi: 10.2147/CCID.S84765. eCollection 2015. PMID 26347269
- [Background] Lin AN, Nakatsui T. Salicylic acid revisited. Int J Dermatol. 1998 May;37(5):335-42. doi: 10.1046/j.1365-4362.1998.00452.x. No abstract available. PMID 9620477
- [Background] Lee HS, Kim IH. Salicylic acid peels for the treatment of acne vulgaris in Asian patients. Dermatol Surg. 2003 Dec;29(12):1196-9; discussion 1199. doi: 10.1111/j.1524-4725.2003.29384.x. PMID 14725662